CLINICAL TRIAL: NCT04880213
Title: A Phase I, Open-label, Single-dose, Sequential Dose Group Study of Orally Administered M5049 Tablet Formulation in Healthy Japanese and Caucasian Participants to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics
Brief Title: Study of M5049 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MS200569_0005; 2020-005408-20 (EudraCT Number)
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Healthy; M5049; Japanese; Caucasian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Japanese: M5049 Dose A (low dose) (Experimental)
  Interventions: Drug: M5049
- Japanese: M5049 Dose B (medium dose) (Experimental)
  Interventions: Drug: M5049
- Japanese: M5049 Dose C (high dose) (Experimental)
  Interventions: Drug: M5049
- Caucasian: M5049 Dose A (low dose) (Experimental)
  Interventions: Drug: M5049
- Caucasian: M5049 Dose B (medium dose) (Experimental)
  Interventions: Drug: M5049
- Caucasian: M5049 Dose C (high dose) (Experimental)
  Interventions: Drug: M5049

INTERVENTIONS:
Drug: M5049 — Participants will receive single oral dose of film-coated tablet M5049 at low dose on Day 1 under fasted condition.
  Arms: Caucasian: M5049 Dose A (low dose); Japanese: M5049 Dose A (low dose)
Drug: M5049 — Participants will receive single oral dose of film-coated tablet M5049 at medium dose on Day 1 under fasted condition.
  Arms: Caucasian: M5049 Dose B (medium dose); Japanese: M5049 Dose B (medium dose)
Drug: M5049 — Participants will receive single oral dose of film-coated tablet M5049 at high dose on Day 1 under fasted condition.
  Arms: Caucasian: M5049 Dose C (high dose); Japanese: M5049 Dose C (high dose)

SUMMARY:
The purpose of this study is to evaluate and determine the safety, tolerability and pharmacokinetics of single-doses of M5049 up to 3 dose levels administered as film-coated tablet under fasted conditions in healthy Japanese and Caucasian participants.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants must be first generation (born in Japan) with both biological parents and all 4 biological grandparents being Japanese native born. Caucasian participants must have both biological parents and 4 biological grandparents of Caucasian descent
* Overtly healthy participants as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring (blood pressure, heart rate and 12-Lead resting ECG)
* Participants with body weight within 45 to 90 kilograms (kg) (female) and 55 to 90 kg (male) and body mass index (BMI) between 18.5 and 29.9 kilograms per meter square (kg/m^2)
* A Caucasian participant will be matched by body weight (± 20% body weight [kg]), height (± 15% height [centimeter (cm) ]) and sex to each Japanese participant
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with history of clinically relevant disease of any organ system that may interfere with the objectives of the study or provide a risk to the health of the participant
* Participants with history of relevant drug hypersensitivity
* Participants with history of splenectomy, epilepsy, other neurological disorders or neuropsychiatric conditions
* Participants with history of a tuberculosis and positive Screening test for hepatitis B surface antigen
* Participants with history of alcoholism or drug abuse
* Other protocol defined exclusion criteria could apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (tlast) (AUC0-tlast) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Area Under Plasma Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC0-inf) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Death | Baseline up to Day 8
Number of Participants with Clinically Significant Changes from Baseline in Laboratory Parameters | Baseline up to Day 3
Number of Participants with Clinically Significant Changes from Baseline in Vital Signs | Baseline up to Day 3
Number of Participants with Clinically Significant Changes from Baseline in 12-lead Electrocardiogram (ECGs) Findings | Baseline up to Day 3

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time Zero to 48 Hours Post-dose (AUC0-48) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Time to Reach Maximum Plasma Concentration (tmax) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Terminal Half-life (t1/2) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Apparent Total Body Clearance (CL/f) of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Apparent Volume of Distribution (Vz/f) During Terminal Phase of M5049 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- [Derived] Klopp-Schulze L, Gopalakrishnan S, Yalkinoglu O, Kuroki Y, Lu H, Goteti K, Krebs-Brown A, Nogueira Filho M, Gradhand U, Fluck M, Shaw J, Dong J, Venkatakrishnan K. Asia-Inclusive Global Development of Enpatoran: Results of an Ethno-Bridging Study, Intrinsic/Extrinsic Factor Assessments and Disease Trajectory Modeling to Inform Design of a Phase II Multiregional Clinical Trial. Clin Pharmacol Ther. 2024 Jun;115(6):1346-1357. doi: 10.1002/cpt.3216. Epub 2024 Feb 28. PMID 38415785
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200569_0005
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html